CLINICAL TRIAL: NCT02452203
Title: Examining the Effects of Reduced Environmental Stimulation on the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Principal Investigator, Justin Feinstein, Principal Investigator, Laureate Institute for Brain Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: float-fMRI-1
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Anxiety
Keywords: floating; interoception
MeSH Terms: conditions — Anxiety Disorders | interventions — Divorce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Floating (Experimental): The participant will float supine in water with a high concentration of Epsom salt for 90 minutes.
  Interventions: Behavioral: Floating
- Chair (Placebo Comparator): The participant will lay in the supine position while reclined in a zero-gravity chair for 90 minutes.
  Interventions: Behavioral: Floating

INTERVENTIONS:
Behavioral: Floating — Floating in either a pool saturated with Epsom salt or in a zero-gravity chair

SUMMARY:
The studies proposed in this protocol aim to explore the anxiolytic properties of floating as it relates to the central and autonomic nervous system.

DETAILED DESCRIPTION:
The human brain is constantly bombarded with sensory information from the external world. This series of studies aim to explore the effects of reducing environmental stimulation using specially designed floatation pools that minimize visual, auditory, tactile, proprioceptive, and thermal input to the brain. Previous research has shown that "floating" in this unique setting can significantly reduce levels of anxiety, stress, blood pressure, and cortisol, while significantly increasing levels of both subjective and physiological forms of relaxation. Much of this past research contained various methodological weaknesses, including small sample sizes, lack of a control group, and no longitudinal follow-up. Moreover, very little is known about the potential benefits of floating in clinical populations, and essentially nothing is known about the effects of floating on the brain. The studies proposed in this protocol aim to further explore floating's potentially salubrious effect on the autonomic nervous system, while beginning to investigate its largely unknown effect on the central nervous system. The researchers have attempted to improve upon the weaknesses of past research by using larger sample sizes, a control group, and a longitudinal design. The current project is focused on documenting the subjective, behavioral, physiological and neural effects of floating in healthy and anxious populations. The subjective effects of floating will be examined using self-report measures and the experience sampling method. The behavioral effects of floating will be examined using measures of interoceptive awareness and distress tolerance. The physiological effects of floating will be examined using waterproof and wireless tracking of blood pressure, heart rate, respiration, and movement, in addition to collecting measures of cortisol and magnesium. A portable electroencephalography (EEG) system will be used to measure sleep during the nights before and after a float experience. The neural effects of floating will be examined using waterproof and wireless EEG collected during the float experience, as well as using functional magnetic resonance imaging (fMRI) collected before and immediately after floating. Using a longitudinal within-subject design, the researchers have a unique opportunity to assess not only functional brain changes, but also structural brain changes induced by repeated exposures to floating. An active control condition aims to control for the effects of simple relaxation by collecting all of the same measures while participants lay supine in a zero-gravity chair situated in a quiet, dimly lit room. This program of research constitutes the first systematic investigation of floating on the body and the brain, and the findings have the potential to illuminate the physiological and neural correlates of the deep relaxation induced by the floating experience.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 18-55 years of age, free of any current or past neurological or psychiatric illness, and capable of performing all tasks during each session of the experiment.
2. They must be able to provide written informed consent and must have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. Participant meets criteria for a DSM5 Axis-1 disorder.
2. Participant endorses current suicidal ideation with intent or plan.
3. Participant fails to adhere to our "Pre-float checklist".
4. Participant is morbidly obese (BMI > 40).
5. Certain drugs or medications consumed within the past week including any psychoactive drugs (e.g., benzodiazepines, opiates, selective serotonin reuptake inhibitors, dopamine agonists, barbiturates, MDMA, LSD, psilocybin, peyote, phencyclidine, ketamine). For all other medications, we require the participant to be stably medicated prior to participation (defined as having taken the medication for 6 weeks or longer).
6. Participant has a history of unstable liver or renal insufficiency; glaucoma; diabetes; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
7. Pregnancy as detected by a urine test.
8. Non-correctable vision or hearing problems.
9. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/ wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Brain activation changes in limbic and paralimbic neural circuitry from pre- to post-float as measured with functional magnetic resonance imaging (fMRI) | fMRI will be undertaken before floating and then immediately following the 3rd float session, an average time frame of 3 weeks
  MRI scan to measure the blood flow changes in the brain

CONTACTS AND LOCATIONS:
Overall Officials: Justin Feinstein, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Zoubi O, Misaki M, Bodurka J, Kuplicki R, Wohlrab C, Schoenhals WA, Refai HH, Khalsa SS, Stein MB, Paulus MP, Feinstein JS. Taking the body off the mind: Decreased functional connectivity between somatomotor and default-mode networks following Floatation-REST. Hum Brain Mapp. 2021 Jul;42(10):3216-3227. doi: 10.1002/hbm.25429. Epub 2021 Apr 9. PMID 33835628